CLINICAL TRIAL: NCT05760456
Title: An Open-label, Randomized, Parallel-controlled Study to Evaluate the Safety and Efficacy of DIDALA Monotherapy in Patients With Type 2 Diabetes Compared With Metformin
Brief Title: Safety and Efficacy of DIDALA Monotherapy in Patients With Type 2 Diabetes Compared With Metformin.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre of Clinical Pharmacology, Hanoi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V5.0 08.08.2022
Record Dates: First submitted 2023-01-30; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DIDALA (Experimental): DIDALA is a herbal medicine, produced from dried mulberry leaves. The drug has been approved by the Drug Administration of Vietnam.
  Interventions: Drug: DIDALA hard capsules
- METFORMIN (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: DIDALA hard capsules — DIDALA is given orally with a dose of 2 capsules, 3 times per day for 12 weeks
  Arms: DIDALA
Drug: Metformin — Metformin 500mg, 1 tablet twice a day, immediately after breakfast and dinner for 12 weeks
  Arms: METFORMIN

SUMMARY:
This is an open-label, two-group parallel study, comparing before and after treatment within the same group and between the two groups. This study is designed to collect data on the safety and efficacy of a marketed pharmaceutical product (DIDALA) compared with Metformin. The efficacy data of DIDALA will be directly compared with Metformin 1000mg/day monotherapy in this study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of enrollment in the study.
* Diagnosed with type 2 diabetes according to the Guidelines for the diagnosis of type 2 diabetes of the Ministry of Health (2011).
* Fasting blood glucose ≤ 10.0 mmol/L.
* No previous treatment with metformin or other antidiabetic drugs.
* Ability and willingness to provide written informed consent and comply with the protocol's requirements.
* Subject who, in the judgment of the Investigator, is likely to be compliant or cooperative during the study.

Exclusion Criteria:

* The patient has been diagnosed with diabetes and has been previously treated with metformin or other antidiabetic agents.
* Patients with indications for insulin therapy or combination therapy of two or more drugs according to the guidelines for diagnosis and treatment of type 2 diabetes of the Ministry of Health.
* Pregnancy or lactation.
* Patients with contraindications to Metformin include severe liver and/or kidney disease, congestive heart failure, cardiovascular collapse, acute myocardial infarction, severe infection, and sepsis.
* Patients with conditions and circumstances that, in the investigator's opinion, are difficult to ensure adherence to study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline at Week 12 in Hemoglobin A1c (HbA1c) | 12 weeks
  Hemoglobin A1c

SECONDARY OUTCOMES:
Change from Baseline at Week 12 in Fasting Plasma Glucose | 12 weeks
  Fasting Plasma Glucose
Safety assessments | 12 weeks
  Safety will be assessed based on the frequency of occurrence of adverse events (AEs) of concern including hypoglycaemic events, clinically significant changes in laboratory parameters (complete blood count, blood biochemistry test), and vital signs during the study period.

CONTACTS AND LOCATIONS:
Locations (2):
- Vietnam (2):
  - Hanoi Hospital of Traditional Medical, Hanoi
  - National Hospital of Traditional Medicine, Hanoi